CLINICAL TRIAL: NCT04180839
Title: Reducing Gaming Cue Reactivity and Behavior Via Retrieval-Extinction Mechanism
Brief Title: Retrieval-extinction Paradigm on Internet Gaming Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R-E_IGD
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gaming-related retrieval-extinction (Experimental): about 30 individuals with IGD will be randomly assigned to the R-E training group
  Interventions: Behavioral: gaming-related retrieval-extinction
- nongaming-related retrieval-extinction (Other): about another 30 individuals with IGD will be randomly assigned to the NR-E training group
  Interventions: Behavioral: nongaming-related retrieval-extinction

INTERVENTIONS:
Behavioral: gaming-related retrieval-extinction — During one training session,participants will first view a 5-min retrieval video containing gaming content and then, 10 minutes later, receive 1-hour of extinction training in which they will be administered four sequences of video, picture and in vivo gaming cues.
  The whole training includes 2 training sessions. Participants will receive one training session once a day for two consectutive days.
  Other Names: R-E
  Arms: gaming-related retrieval-extinction
Behavioral: nongaming-related retrieval-extinction — During one session,participants will first view a 5-min neutral video and then, 10 minutes later, receive 1-hour of extinction training in which they will be administered four sequences of video, picture and in vivo gaming cues.
  The whole procedure includes 2 sessions. Participants will receive one session once a day for two consectutive days.
  Other Names: NR-E
  Arms: nongaming-related retrieval-extinction

SUMMARY:
The overall aim of this experimental study is to apply the new paradigm of substance addiction intervention to the study of Internet gaming disorder(IGD) subjects' intervention.

DETAILED DESCRIPTION:
This study is based on the retrieval-extinction paradigm.As with the efficacy, the experiment aims to test the effect of the retrieval-extinction paradigm on game craving and behave of IGD subjects, so as to provide an empirical basis for the development of effective intervention means of Internet gaming disorder.

ELIGIBILITY:
Inclusion Criteria:

1. the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5 ) recommended diagnosis of Internet gaming disorder : the scores of the 9 items of DSM-5 recommended diagnosis for Internet gaming disorder ≥ 5.
2. the scores of the Young-Internet addiction Test ≥ 50
3. engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.

Exclusion Criteria:

1. current or history of use of illegal substances and other addictions;
2. current or history of psychiatric or neurological illness;
3. current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in gaming craving at cue-reactivity task between the two test sessions | baseline , one day after training
  Participants were asked to passively watch three kinds of videos and rate their craving immediately after each video clip using 10-point visual analog scales.The task assesses the severity of cue-induced craving for Internet gaming, with high scores indicating great cue-induced craving.

SECONDARY OUTCOMES:
Mean Change in gaming Craving | The questionnaire is given to participants to record their gaming craving at baseline、after the first day of training、after the second day of training、one day after training、1 week and 1 month after tranning respectively
  The Brief Questionnaire of gaming Urges questionnaire is a 10-item gaming urge questionnaire with scores ranging from 0 to 10 to assess gaming craving. The questionnaire assesses the severity of craving for Internet gaming behavior, with high scores indicating great craving.
Mean Change in gaming time at baseline、1-Week and 1-month Follow-Up | A diary is given to participants to record their gaming time at baseline、 1-week and 1-month
  At the baseline、end of the first week and month test session, participants will receive a diary in which to record the gaming time after the 1-week and 1-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: jintao Zhang, phD, Principal Investigator — Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
we will share individual participant data when required
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after the publication of related paper , for 3 years
Access Criteria: By contacting the principal investigator. Email : zhangjintao@bnu.edu.cn

REFERENCES:
- [Background] Xue YX, Luo YX, Wu P, Shi HS, Xue LF, Chen C, Zhu WL, Ding ZB, Bao YP, Shi J, Epstein DH, Shaham Y, Lu L. A memory retrieval-extinction procedure to prevent drug craving and relapse. Science. 2012 Apr 13;336(6078):241-5. doi: 10.1126/science.1215070. PMID 22499948